CLINICAL TRIAL: NCT01209156
Title: A Phase 1 Evaluation of the Kinetics, Clearance and Cerebral Distribution of One Novel PBR PET Imaging Agent, 18F-PBR-111 Following Intravenous Administration in Healthy Subjects and Alzheimer Disease Patients
Brief Title: Evaluation of [18F] PBR111 and PET as a Marker of Inflammation in Subjects With Neurological Conditions
Acronym: PBR111
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, Danna Jennings, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PBR111 001
Record Dates: First submitted 2010-09-20; First posted 2010-09-27 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 2-(6-chloro-2-(4-(3-fluoropropoxy)phenyl)imidazo(1,2-a)pyridin-3-yl)-N,N-diethylacetamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Assess [18F] PBR111 and PET imaging (Experimental): Evaluation of PET imaging with [18F]PBR111 in HV and AD subjects (Proof of Mechanism)
  Interventions: Drug: [18F] PBR111

INTERVENTIONS:
Drug: [18F] PBR111 — Subjects will be injected with 5mCi (not to exceed a maximum of 5.5 mCi) of [18F]PBR111, followed by PET imaging.

SUMMARY:
The underlying goal of this study is to assess PBR-111 positron emission tomography (PET) imaging as a tool to detect microglial activation in the brain of Alzheimer disease (AD) research participants and age- and gender-matched healthy volunteers.

DETAILED DESCRIPTION:
This is a phase 1, open-label, single-center, non-randomized single dose study to assess the kinetics, clearance and cerebral distribution of PBR-111 positron emission tomography (PET) imaging in detecting microglial activation in the brain in patients with probable Alzheimer disease (AD) compared to healthy volunteers (HVs). All aspects related to image acquisition, processing and visual as well as quantitative evaluation will be developed, optimized and validated (where required).

Each subject will be required to visit the study center during the screening phase and on the PBR-111 PET imaging day (baseline). A telephone follow-up visit will be performed 7 days (+/- 3 days) after PBR-111 PET administration.

At the screening visit, each subject (or caregiver in the case of AD subjects) will be asked to provide written informed consent or assent. During the screening phase (maximum duration - 60 days) subject medical, neurological and surgical history, clinical assessments and a neuro-psychiatric evaluation will be performed on all eligible subjects. Subjects will be allowed to leave the center after all evaluations have been completed. During this period an MRI of the brain will be performed. During the PBR-111 PET imaging day, all subjects will receive a single IV injection of PBR-111 and scanning will be performed over a 3.5 hour period. Each subject will have a telephone follow-up 7 days (+/- 3 days) thereafter to assess for adverse events.

ELIGIBILITY:
INCLUSION CRITERIA: Alzheimer Disease (AD)

1. The participant is 50 years or older.
2. Written informed consent is obtained.
3. Participants have a clinical diagnosis of probable Alzheimer disease based on National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer Disease and Related Disorders Association (NINCDS/ADRDA) criteria.
4. Does not fulfill the ICC criteria for probable DLB (Appendix 3), the NINDS-AIREN for probable Vascular dementia (Appendix 5), or the Neary [Neary et al. 1998] criteria for FTD (Appendix 4)
5. Clinical Dementia Rating Scale score ≤ 2.
6. Modified Hachinski Ischemia Scale score of ≤ 4.
7. MRI brain scan findings that do not reveal changes indicative of stroke and/or generalized cerebrovascular disease (e.g., the ARWMC scale) changes limited to: a white matter lesion score of 0 or 1 or 2 and a basal ganglia score of 0 or 1)
8. has a caregiver willing and able to attend all study visits and perform the psychometric tests requiring the presence of a caregiver
9. For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-PBR111 injection.

EXCLUSION CRITERIA: Alzheimer Disease (AD)

1. History of significant cerebrovascular disease.
2. Clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
3. Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
4. Pregnancy
5. Contraindication to MRI examination, e.g. metal implants or phobia as determined by the onsite radiologist performing the scan
6. History of exposure to any radiation >15 mSv/year (e.g. occupational or radiation therapy)
7. Receiving drug therapy or other treatment that is known to lead to greatly fluctuating values of the hematological or chemical laboratory parameters or to severe side effects (e.g. chemotherapy)
8. Received anti-amyloid drug therapy.

INCLUSION CRITERIA: Healthy Volunteer (HV)

1. The participant is 18 years or older, with at least 4 subjects ≥50 years.
2. Written informed consent is obtained.
3. Negative history of neurological or psychiatric illness based on evaluation by a research physician.
4. Has no evidence of cognitive impairment as indicated by a clinical dementia rating (CDR, [Hughes et al. 1993]) score of 0 (zero) and a score of ≥ 28 in the Mini-Mental Status Examination (MMSE, [Folstein et al. 1975]) Clinical Dementia Rating score = 0.
5. has MRI brain scan that has been judged as "normal (age- appropriate)" including ARWMC scale [Wahlund et al. 2001] scores supporting the lack of cerebrovascular disease (e.g., a white matter lesion score of 0 or 1 or 2 and a basal ganglia score of 0 or 1) and a Scheltens scale [Scheltens et al. 1992] verifying the lack of cerebral atrophy (e.g. bilateral temporal lobe atrophy visual score of 0 or 1)
6. For females, non-child bearing potential a negative urine or blood pregnancy test on day of [18F]-PBR-111 injection.

EXCLUSION CRITERIA: Healthy Volunteer (HV)

1. History of significant cerebrovascular disease.
2. Clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
3. Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
4. Pregnancy
5. Contraindication to MRI examination, e.g. metal implants or phobia as determined by the on-site radiologist performing the scan
6. History of exposure to any radiation >15 mSv/year (e.g. occupational or radiation therapy)
7. Receiving drug therapy or other treatment that is known to lead to greatly fluctuating values of the hematological or chemical laboratory parameters or to severe side effects (e.g. chemotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the cerebral distribution of [18F]PBR-111 positron emission tomography (PET) for detection/exclusion of microglial activation in patients with Alzheimer Disease compared to healthy volunteers. | 1 year

SECONDARY OUTCOMES:
To assess the dynamic uptake and washout of [18F]PBR-111, a potential imaging biomarker for inflammatory changes in brain, using positron emission tomography (PET) in Alzheimer disease subjects compared to healthy volunteers. | 1 year
To perform blood metabolite characterization of [18F]PBR-111 in AD subjects compared to Healthy volunteers to determine the nature of metabolites in assessment of [18F]PBR-111 as a single positron computed tomography (PET) brain imaging agent. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States